CLINICAL TRIAL: NCT00566787
Title: A Prospective, Multi-center Study With Case Matched Controls to Evaluate the Safety and Efficacy of the AtriCure Bipolar System for the Treatment of Continuous Atrial Fibrillation as Adjunct Therapy to Elective Open Heart Surgery
Brief Title: Concomitant Treatment of Permanent Atrial Fibrillation
Acronym: RESTORE SR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2003-1
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Atrial Fibrillation
Keywords: AF; Atrial Fibrillation; afib; racing heart; cabg; valve; ablation; bipolar; radiofrequency; rf
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia

INTERVENTIONS:
Device: Surgical bipolar radiofrequency ablation using the AtriCure Bipolar System — Surgical bipolar radiofrequency ablation using the AtriCure Bipolar System

SUMMARY:
RESTORE-SR study is a multi-center, prospective, nonrandomized study with case matched concurrent controls to evaluate the safety and efficacy of the AtriCure Bipolar System

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subject between 18 to 80 years of age
2. Subject is scheduled to undergo elective cardiac surgical procedure(s) to be performed on cardiopulmonary bypass including:

   * coronary artery bypass and/or
   * mitral valve surgery (repair or replacement)
   * aortic valve surgery (repair or replacement)
   * tricuspid valve surgery (repair or replacement)
3. Left Ventricular Ejection Fraction ≥ 30%
4. Subject is willing and able to provide written informed consent
5. Subject has a life expectancy of at least 2 years
6. Subject is willing and able to return for scheduled follow-up visits
7. TREATMENT SUBJECTS ONLY: Subject has a 3 month documented history of continuous atrial fibrillation
8. CONTROL SUBJECTS ONLY: Subject is not in atrial fibrillation at time of surgery

Exclusion Criteria:

1. Lone AF without indication(s) for concomitant CABG and/or mitral valve surgery, aortic valve surgery, tricuspid valve surgery or double valve surgery
2. Prior cardiac surgery (Redo -including previous ablation)
3. Patient requires atrial septal defect repair or any other concomitant open-heart procedure, other than CABG and/or mitral valve surgery; aortic valve surgery, tricuspid valve surgery or double valve surgery
4. Serum creatinine concentration greater than 2.0 mg/dl
5. Class IV NYHA heart failure symptoms and/or Class IV CCS anginal symptoms
6. Prior history of cerebrovascular accident within 6 months or at any time if there is residual neurologic deficit
7. Active infection
8. Known carotid artery stenosis greater than 80%
9. Severe peripheral arterial occlusive disease defined as claudication with minimal exertion
10. A known drug and/or alcohol addiction
11. Mental impairment or other conditions which may not allow the the subject to understand the nature, significance and scope of the study
12. Pregnancy or desire to get pregnant within 12 months of study enrollment
13. Requires anti-arrhythmic drug therapy for the treatment of a ventricular arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint is the proportion of treated patients who are free of atrial fibrillation without the need for anti-arrhythmic agents at the six-month follow-up visit. | 6 months
The primary safety endpoint is the occurrence of serious adverse events that are considered to be associated with the Maze procedure. | 30 days

SECONDARY OUTCOMES:
The secondary efficacy endpoint is the proportion of patients in the treatment group who are free of atrial fibrillation independent of the need for anti-arrhythmic drugs. | 6 Months
The secondary safety endpoints are: total cross clamp time, total time on bypass, length of hospital stay (days), and length of ICU stay (hours) | Discharge

CONTACTS AND LOCATIONS:
Overall Officials: A. Marc Gillinov, MD, Principal Investigator — The Cleveland Clinic
Locations (10):
- United States (10):
  - Heart Center of Indiana, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - The Methodist Hospital, Houston, Texas
  - Sentara Norfolk Hospital, Norfolk, Virginia
  - Sacred Heart Medical Center, Seattle, Washington
  - St. Mary's Hospital Medical Center, Madison, Wisconsin